CLINICAL TRIAL: NCT03978676
Title: Exercise-induced in Secondary Mitral Regurgitation: Analysis of Echocardiographic Parameters at Rest Predicting the Onset of Significant Exercise-induced Mitral Regurgitation
Acronym: IM EFFORT
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IM EFFORT
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Secondary mitral insufficiency is a common complication of heart failure, aggravating symptoms and prognosis, and may be responsible for worsening dyspnea, pulmonary edema, and excess mortality. It is essentially a ventricular rather than a valvular disease, whose origin may be ischemic or not. It is induced by a geometrical and contractile modification of the left ventricle which causes an imbalance between the tensile and the closing forces of the mitral valve thus causing a defect of coaptation and the increase of the surface between the mitral leaves and the ring in systole (tenting). Dynamic mitral insufficiency is defined by changes in the degree of severity of regurgitation as a function of hemodynamic conditions.

During exercise, the course of mitral insufficiency is variable and is not predicted by the degree of regurgitation at rest. The worsening of the leak is also well correlated with the onset of dyspnea on exertion in patients with left Ventricular Ejection Fraction heart failure (LVEF reduced). Nevertheless, there is little data available in the literature on the factors predisposing to the development of stress-related mitral insufficiency, as well as its clinical and echocardiographic impact in the cardiac insufficiency patient, particularly in the case of preserved LVEF (6.7%).

The identification of echocardiographic data at rest to predict and anticipate the behavior of mitral insufficiency in the effort (aggravation or stability / disappearance), would allow a simplified evaluation and a better management in this population of patients for which the evaluation in echography of effort can be technically complex and limited (difficulty of quantification of the mitral leak, time of effort sometimes too short ...).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient who received a stress echocardiography performed by an experienced operator in the evaluation of mitral insufficiency at the Paris Saint-Joseph Hospital Group between March 2016 and February 2019
* Patient presenting during this ultrasound a mitral insufficiency secondary to rest and effort
* Francophone patient

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients who oppose the use of their data for this research
* Patient with primary mitral insufficiency, structural abnormality of valvular leaflets
* Patient with valvular or valvular calcification
* Patient with other significant associated valvulopathy (grade> II / IV: corresponds to the severity of mitral leak quantified on cardiac ultrasound)
* Patient with cardiac valve prosthesis
* Hypertrophic or restrictive cardiomyopathy
* Patient with congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who received a stress echocardiography performed by an experienced operator in the evaluation of mitral insufficiency at the Paris Saint-Joseph Hospital Group between March 2016 and February 2019 and presenting during this ultrasound a mitral insufficiency secondary to rest and effort
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Aggravation of secondary mitral insuffiency | Day 1
  Il will measure an increase of the grade of severity of at least 1/4 compared to the rest.
Aggravation of secondary mitral insuffiency | Day 1
  Il will measure an increase of the ORS of more than 0.5 cm² in case of IM Grade 4 at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Garçon, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France